CLINICAL TRIAL: NCT00105911
Title: A Cognitive-Behavioral Intervention for Depression and Anxiety in COPD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IIR 00-097
Record Dates: First submitted 2005-03-17; First posted 2005-03-18 (Estimated); Last update posted 2015-04-07 (Estimated); Status verified 2007-02

CONDITIONS: Depressive Disorders; Anxiety Disorders; Pulmonary Disease, Chronic Obstructive
Keywords: Cognitive Behavioral Therapy
MeSH Terms: conditions — Depressive Disorder; Anxiety Disorders; Pulmonary Disease, Chronic Obstructive | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm 1 (Other)
  Interventions: Behavioral: Cognitive Behavioral Therapy

INTERVENTIONS:
Behavioral: Cognitive Behavioral Therapy

SUMMARY:
The literature and our preliminary studies found that in COPD patients, psychosocial factors affect quality of life (QOL) and functioning more than would be expected given the severity of their disease. To improve QOL and functioning in the approximately 50% of COPD patients with significant anxiety and/or depressive symptoms, interventions are needed. Much research documents the utility of cognitive behavioral therapy (CBT) in treating depression and anxiety, showing it to have promise as a self-management intervention to improve QOL in COPD patients.

DETAILED DESCRIPTION:
Background:

The literature and our preliminary studies found that in COPD patients, psychosocial factors affect quality of life (QOL) and functioning more than would be expected given the severity of their disease. To improve QOL and functioning in the approximately 50% of COPD patients with significant anxiety and/or depressive symptoms, interventions are needed. Much research documents the utility of cognitive behavioral therapy (CBT) in treating depression and anxiety, showing it to have promise as a self-management intervention to improve QOL in COPD patients.

Objectives:

Objectives were to compare CBT for anxiety and depression with COPD education for COPD patients with moderate-to-severe anxiety and/or depressive symptoms.

Methods:

Veterans were recruited from VAMC clinics and through press releases. Two hundred and thirty-eight COPD patients with comorbid anxiety and/or depressive symptoms were randomized to either 8 weeks of CBT/usual care or 8 weeks of COPD Education/usual care. We hypothesized that COPD patients receiving CBT/usual care would improve more than COPD patients receiving COPD Education/usual care. Improvement was defined as increased disease-specific QOL, generic QOL, and 6-minute walk distance; and decreased depression, anxiety, and health service use. Outcomes were examined pre-, mid- and post-treatment and at 4, 8 and 12 months.

Status:

The study was scheduled to officially end December 31, 2005, but was granted a no-cost extension by HSR&D to complete data analyses and prepare final papers. The extension was granted through June 30, 2006. As of the date of this final report, the study is complete.

ELIGIBILITY:
Inclusion Criteria:

Moderate depression or anxiety, COPD

Exclusion Criteria:

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 222 (Estimated)
Dates: Start 2002-07; Study Completion 2005-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark E. Kunik, MD MPH, Principal Investigator — Michael E. DeBakey VA Medical Center, Houston, TX
Locations (1):
- Michael E. DeBakey VA Medical Center, Houston, TX, Houston, Texas, United States

REFERENCES:
- [Result] Maurer J, Rebbapragada V, Borson S, Goldstein R, Kunik ME, Yohannes AM, Hanania NA; ACCP Workshop Panel on Anxiety and Depression in COPD. Anxiety and depression in COPD: current understanding, unanswered questions, and research needs. Chest. 2008 Oct;134(4 Suppl):43S-56S. doi: 10.1378/chest.08-0342. PMID 18842932
- [Result] Kunik ME, Veazey C, Cully JA, Souchek J, Graham DP, Hopko D, Carter R, Sharafkhaneh A, Goepfert EJ, Wray N, Stanley MA. COPD education and cognitive behavioral therapy group treatment for clinically significant symptoms of depression and anxiety in COPD patients: a randomized controlled trial. Psychol Med. 2008 Mar;38(3):385-96. doi: 10.1017/S0033291707001687. Epub 2007 Oct 9. PMID 17922939
- [Result] Kunik ME, Azzam PN, Souchek J, Cully JA, Wray NP, Krishnan LL, Nelson HA, Stanley MA. A practical screening tool for anxiety and depression in patients with chronic breathing disorders. Psychosomatics. 2007 Jan-Feb;48(1):16-21. doi: 10.1176/appi.psy.48.1.16. PMID 17209145
- [Result] Cully JA, Graham DP, Stanley MA, Kunik ME. Depressed and Anxious COPD Patients: Predictors of Psychotherapy Engagement from a Clinical Trial. Journal of Clinical Psychology in Medical Settings. 2007 Jan 1; 14:160-164.
- [Result] Kraus CA, Kunik ME, Stanley MA. Use of cognitive behavioral therapy in late-life psychiatric disorders. Geriatrics. 2007 Jun;62(6):21-6. PMID 17547480
- [Result] Burgess A, Kunik ME, Stanley MA. Chronic obstructive pulmonary disease: assessing and treating psychological issues in patients with COPD. Geriatrics. 2005 Dec;60(12):18-21. No abstract available. PMID 16343032
- [Result] Roundy K, Cully JA, Stanley MA, Veazey C, Souchek J, Wray NP, Kunik ME. Are anxiety and depression addressed in primary care patients with chronic obstructive pulmonary disease? A chart review. Prim Care Companion J Clin Psychiatry. 2005;7(5):213-8. doi: 10.4088/pcc.v07n0501. PMID 16308576
- [Result] Kunik ME, Roundy K, Veazey C, Souchek J, Richardson P, Wray NP, Stanley MA. Surprisingly high prevalence of anxiety and depression in chronic breathing disorders. Chest. 2005 Apr;127(4):1205-11. doi: 10.1378/chest.127.4.1205. PMID 15821196
- [Result] Stanley MA, Veazey C, Hopko D, Diefenback G, Kunik ME. Anxiety and Depression in chronic obstructive pulmonary disease: a new intervention and case report. Cognitive and behavioral practice. 2005 Dec 1; 12(4):424-436.
- [Result] Cully JA, Graham DP, Stanley MA, Ferguson CJ, Sharafkhaneh A, Souchek J, Kunik ME. Quality of life in patients with chronic obstructive pulmonary disease and comorbid anxiety or depression. Psychosomatics. 2006 Jul-Aug;47(4):312-9. doi: 10.1176/appi.psy.47.4.312. PMID 16844889
- [Result] Ferguson CJ, Stanley M, Souchek J, Kunik ME. The utility of somatic symptoms as indicators of depression and anxiety in military veterans with chronic obstructive pulmonary disease. Depress Anxiety. 2006;23(1):42-9. doi: 10.1002/da.20136. PMID 16315269